CLINICAL TRIAL: NCT04243876
Title: Comparison of the Relationship Between Age and Serum Paraoxonase /Arylesterase Activity of Patients With Acute Coronary Syndrome Presenting to the Emergency Department''
Brief Title: Decrease in Paraoxonase Enzyme Level and Myocardial İnfarction
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Bahadir Taslidere, Associate Professor, clinical research, Bezmialem Vakif University
Other Study IDs: 20/9
Record Dates: First submitted 2019-12-31; First posted 2020-01-28 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Myocardial Infarction; High-Density Lipoid Deficiency
Keywords: Myocardial infarction, Paraoxonase
MeSH Terms: conditions — Myocardial Infarction; Hypoalphalipoproteinemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- paraoxanase: Enzyme level
  Interventions: Diagnostic Test: paraoxanase enzyme level
- Myocardial infarction: RESULTS OF ANGIOGRAPHY
  Interventions: Diagnostic Test: paraoxanase enzyme level

INTERVENTIONS:
Diagnostic Test: paraoxanase enzyme level — presence of paraoxonase enzyme deficiency and associated troponin elevation
  Other Names: troponin level; HDL level

SUMMARY:
Myocardial infarction is a polygenic disease that may occur due to various environmental risk factors. Mortality risk of the disease; sex, age, smoking, systolic blood pressure, total cholesterol, and high-density lipoprotein levels. The paraoxonase-1 phenotype is expressed as the paraoxonase/arylesterase ratio and is closely related to high-density lipoprotein, acting as an endogenous defense mechanism against vascular oxidative stress, thus contributing to the prevention of atherosclerosis. Serum concentration and activity depend on environmental factors as well as genetic polymorphism. This decrease in enzyme concentration causes changes in gene expression (1). Numerous data on Paraoxonase-1 levels have been found in studies, especially with decreasing serum paraoxonase and arylesterase activities with age, associated with increased risk of systemic oxidative stress and atherosclerosis in humans. Many studies have shown that serum Paraoxonase-1 activity is significantly reduced in people with myocardial infarction, dyslipidemia, atherosclerosis, and chronic kidney disease. The most important risk factor for these and similar diseases is aging. Diversity of conditions such as genetic predisposition, malnutrition, stress, and smoking, which increases vascular dysfunction due to oxidative stress, classify individuals with acute myocardial infarction according to age groups and investigate whether there is a relationship between serum Paraoxonase-1 activity and severity of coronary artery disease in young patients. The paraoxonase-1 enzyme, which is known to decrease blood levels with age, is found to be significantly lower in patients with myocardial infarction at a young age compared to the healthy control group.

DETAILED DESCRIPTION:
High-density lipoprotein (HDL), known as good cholesterol, is named because of its protective effects on the cardiovascular system. in order to summarize the mechanism of the event, cholesterol is transported from the liver to the cells and from the cells back to the liver via blood. Cholesterol and other fats are carried in packets called lipoprotein to dissolve in the blood. Those with these are two kinds of cholesterol, these low-density lipoproteins and good cholesterol can help to lower the cholesterol as well. LDL cholesterol is the main package that carries cholesterol in the blood. When the blood is high, it sticks to the inside of the veins and forms plaques around here. With the addition of cholesterol, a blood clot that formed in cracks that occur on these plaques grow the arteries and clogs them. If the blockage occurs in the heart vessels, it can cause a heart attack and stroke. Cholesterol in the blood is a part of a package called HDL-cholesterol is carried in. HDL-cholesterol prevents the accumulation of cholesterol in the veins.

It collects the cholesterol circulating in the blood and brings it to the liver to get rid of it from the body. Thus, it reduces the exposure of blood vessels to the harmful effects of cholesterol. All these effects of HDL cholesterol in the paraoxonase enzyme owes. This may be the reason why Dolat may even use another nomenclature instead of HDL in future years. A paraoxonase-1 enzyme, which is known to decrease blood level with age, is found to be significantly lower in patients with myocardial infarction at a young age compared with the healthy control group in this study, and the measurement of this enzyme level can be used as a screening test in people with risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18
* All acute coronary syndrome patients

Exclusion Criteria:

- Patients with normal angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the emergency department over the age of 18
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
early diagnosis | one year
  paraoxonase enzyme measurement

CONTACTS AND LOCATIONS:
Overall Officials: bahadir taslidere, Principal Investigator — BEZMİALEM VAKİF UNİVERSİTY
Locations (1):
- Bezmialem vakif university, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
nope

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04243876/Prot_SAP_ICF_000.pdf